CLINICAL TRIAL: NCT06018077
Title: Investıgatıon of The Relatıonshıps Between Serum Chemerın Levels, Dıet Qualıty, Inflammatory and Phytochemıcal Indıces in Adults wıth Colorectal Cancer
Brief Title: Chemerin in Colorectal Cancer and Its Relationship With Diet Quality
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Collaborators: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Semra Bakir Angay, Principal Investigator, Hacettepe University
Other Study IDs: GO22/297
Record Dates: First submitted 2023-08-25; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer; Diet, Healthy; Diet Habit; Nutrition Aspect of Cancer; Inflammation
Keywords: Colorectal cancer; Dietary inflammatory index; Dietary phytochemical index; Chemerin; Dietary total antioxidant capacity
MeSH Terms: conditions — Colorectal Neoplasms; Feeding Behavior; Inflammation | interventions — Eating; Diet Records; Blood Specimen Collection; Weights and Measures; Body Height; Basal Metabolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — 1 tube of blood sample is centrifuged and serum is taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colorectal Cancer Group: Individuals aged 18-65 years, who applied to Ankara City Hospital Oncology Hospital Medical Oncology Outpatient Clinic, newly diagnosed with colorectal cancer as a result of the necessary examinations, at least 3 weeks after the surgical procedure and without metastasis (except for Stage IV)
  Interventions: Behavioral: Dietary İntake, Biochemical parameters, Antropometric measuruments
- Healthy Group: A healthy adult between the ages of 18-65 who has not been diagnosed with any malignant disease and consented to participate in the study.
  Interventions: Behavioral: Dietary İntake, Biochemical parameters, Antropometric measuruments

INTERVENTIONS:
Behavioral: Dietary İntake, Biochemical parameters, Antropometric measuruments — Nutritional status of individuals will be evaluated with a 24-hour retrospective food consumption record and food consumption frequency questionnaire. After 8-12 hours of fasting, body composition analysis will be performed and within the scope of anthropometric measurements, body weight, height length, BMI measurements will be taken. Then, venous blood will be taken from the participants C-reactive protein (CRP), albumin and chemerin level will be analyzed.
  Other Names: Food Frequency Questionnaire and Dietary Record; Blood Sample; Antropometric measurements (body weight, height, body fat rate, muscle rate, resting metabolic rate)

SUMMARY:
To investigate the relationship between serum chemerin levels of individuals with colorectal cancer and systematic inflammatory response parameters such as C-reactive protein(CRP) and albumin, and to investigate the relationship of these biomarkers with dietary inflammatory index, phytochemical, anthropometric measurements, and dietary inflammatory index, which is calculated with the data obtained from the 24-hour food consumption record and food consumption frequency questionnaire. The aim of this study is to examine the relationships between the index and dietary antioxidant capacity and to compare them with those of healthy individuals.

DETAILED DESCRIPTION:
The research will be executed. with 52 adult individuals between the ages of 18-65 who applied to the Ankara City Hospital Oncology Hospital Medical Oncology outpatient clinic, newly diagnosed with colorectal cancer (except for Stage IV), and 52 healthy adult individuals without any chronic disease, matched for age, gender, and BMI. Individuals will be told about the study in detail and those who accept will be included in the study by signing an informed consent form. A data collection form containing health and demographic information will be applied to the participants; Then, after 8-12 hours of fasting, body composition analysis (body fat ratio, muscle ratio, visceral fat level, resting metabolic rate) will be performed with the Omron BF511, a body composition analysis scale that works with the bioelectrical impedance method, and within the scope of anthropometric measurements, body weight, height length, BMI measurements will be taken. Body mass index (BMI) will be obtained by dividing the body weight (kg) by the square of the height in meters. After 8-12 hours of fasting, 5 ml of venous blood will be taken from the participants by the nurses of the Medical Oncology Clinic, and the serum obtained after centrifugation will be analyzed in accordance with the manufacturer's kit protocols and in duplicate, the C-reactive protein (CRP) level will be analyzed by the immunoturbidimetric method and the albumin Bromocresol Green-Dye binding method, and chemerin level by enzyme-linked immunoassay (ELISA) method. Nutritional status of individuals will be evaluated with a 24-hour retrospective food consumption record and food consumption frequency questionnaire, and dietary inflammatory index, phytochemical index, and dietary antioxidant capacity will be calculated from the obtained records. In order to measure the inflammatory potential of the diet, the Dietary Inflammatory Index (DII) was developed based on the pro-inflammatory and anti-inflammatory effects of different dietary components on various inflammatory biomarkers. The "Phytochemical Index" method was used to calculate the total phytochemical intake from the diet. The total antioxidant capacity of the diet was calculated using data obtained from dietary intake records based on Ferric Reducing Ability of Plasma (FRAP) methods.

ELIGIBILITY:
Inclusion Criteria:

For patient group

* Between the ages of 18-65,
* At least 3 weeks after surgery
* Individuals newly diagnosed with colorectal cancer by a oncolog (except for Stage IV)

For healthy group

* Between the ages of 18-65,
* Healthy adult individuals without any chronic disease

Exclusion Criteria:

For patient group

* Receiving active radiotherapy or chemotherapy,
* Existing history of metastasis,
* Having a malignant disease other than the diagnosis of colorectal cancer, - History of metabolic syndrome, cardiovascular disease, hepatic disease, chronic kidney disease, major hormonal or hematological disease, pulmonary disease,
* With a history of autoimmune disease, with a history of inflammatory diseases (pancreatitis, chron's, ulcerative colitis, etc.),
* Those who use nonsteroidal anti-inflammatory drugs (NSAIDs),
* Alcoholic and other drug addicts,
* Smokers,
* Those with mental disorders (major depressive disorder, dementia),
* Those who take corticosteroid or hormone therapy,
* Those who have an existing infectious disease, those who receive medical nutrition therapy for any disease

For healthy group

* Individuals aged 18 and under and 65 years and older,
* History of metabolic syndrome, cardiovascular disease, hepatic disease, chronic kidney disease, major hormonal or hematological disease, pulmonary disease,
* With a history of autoimmune disease, with a history of inflammatory diseases (pancreatitis, chron's, ulcerative colitis, etc.),
* Those who use nonsteroidal anti-inflammatory drugs (NSAIDs),
* Pregnant and lactating women,
* Alcoholic and other drug addicts,
* Smokers, those with mental disorders (major depressive disorder, dementia),
* Those taking corticosteroid or hormone therapy,
* Those with existing infectious disease,
* Those receiving medical nutrition therapy for any illness

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: After the necessary tests are made by the doctor of Ankara City Hospital Oncology Hospital Medical Oncology Polyclinic, individuals diagnosed as colorectal in the patient group, and those evaluated as healthy in the control group and meet the eligibility criteria will be included.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Serum chemerin level | 12 months
  The blood obtained from individuals after 8-12 hours of fasting will be analyzed in duplicate with the enzyme-linked immunity test (ELISA) method from the serum obtained after centrifugation, in accordance with the manufacturer's kit protocols.
Body weight | 12 months
  The body weights of the individuals will be measured after 8-12 hours of fasting, using Omron BF511 brand bioelectrical impedance device, wearing light clothes without metal objects.
Body fat percentage | 12 months
  The body fat percentage of the individuals will be measured after 8-12 hours of fasting, using Omron BF511 brand bioelectrical impedance device, wearing light clothes without metal objects.
Body muscle percentage | 12 months
  The body muscle percentage of the individuals will be measured after 8-12 hours of fasting, using Omron BF511 brand bioelectrical impedance device, wearing light clothes without metal objects.
Visseral fat level | 12 months
  The visseral fat level of the individuals will be measured by using Omron BF511 brand bioelectrical impedance device while they are on an empty stomach and wearing light clothes without metal objects.
Serum albumin level | 12 months
  The blood obtained from individuals after 8-12 hours of fasting will be analyzed from the serum obtained after centrifugation, in duplicate using the Bromocresol Green-Dye binding method, in accordance with the manufacturer's kit protocols.
Serum C-reaktive protein (CRP) | 12 months
  The blood obtained from individuals after 8-12 hours of fasting will be analyzed in duplicate with the immunoturbidimetric method from the serum obtained after centrifugation, in accordance with the manufacturer's kit protocols.
Body Mass Index (BMI) | 12 months
  Body mass index (BMI) will be obtained by dividing the body weight (kg) by the square of the height in meters.
Resting Metabolic Rate (RMR) | 12 months
  The resting metabolic rate of the individuals will be measured by using Omron BF511 brand bioelectrical impedance device while they are on an empty stomach and wearing light clothes without metal objects.
Dietary Phytochemical Index (DPI) | 12 months
  he "Phytochemical Index" method was used to calculate the total phytochemical intake from the diet. The ratio of the total amount of phytochemical rich foods in the diet in grams per day to the total food intake (g/day) will be calculated as follows. The amount of phytochemicals contained in each food will be obtained from the USDA database.
Dietary Inflammatory Index (DII) | 12 months
  The frequency of food consumption from the participants and the data to be obtained from the twenty-four hour retrospective food consumption record will be evaluated using the Computer Aided Nutrition Program Nutrition Information System (BeBIS 9.0). "Diet inflammatory index" will be calculated by multiplying the nutritional parameters obtained from the recordings with the "inflammatory effect score".The resulting values are summed to obtain the dietary inflammatory index (DII) score, which represents the inflammatory load of the individual's daily diet.
Dİetary Total Antioxidant Capacity (DTAC) | 12 months
  Dietary total antioxidant capacity will be determined using the 'Antioxidant Food Database'. The FRAP value of that food will be calculated by multiplying the reported iron reducing antioxidant power (FRAP) value for each food and the grams of the daily average consumed food. The total antioxidant capacity (TAK) of the diet will be calculated by summing the calculated FRAP values of all foods and expressed as mmol/100 g nutrient.

CONTACTS AND LOCATIONS:
Overall Officials: Semra Bakir Angay, Principal Investigator — Hacettepe University; Aylin Acikgoz Pinar, Principal Investigator — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University Health Science Faculty, Nutrition and Dietetic Department, Ankara
  - Ankara Bilkent City Hospital, Oncology Hospital, Medical Oncology Outpatient Clinic, Ankara